CLINICAL TRIAL: NCT02424734
Title: Open-label, Multicentre Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Efficacy Of Ceftaroline In Neonates And Young Infants With Late-onset Sepsis
Brief Title: Safety, Tolerability and Efficacy of Ceftaroline in Paediatrics With Late-Onset Sepsis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated on 22Dec2017 due to slow enrollment; there were no safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: D3720C00009; C2661002 (Other: Alias Study Number); 2014-003243-34 (EudraCT Number)
Record Dates: First submitted 2015-02-23; First posted 2015-04-23 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Late-onset Sepsis
Keywords: Late-onset Sepsis
MeSH Terms: interventions — Ceftaroline; Ampicillin; Aminoglycosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceftaroline Fosamil (Experimental): Ceftaroline Fosamil
  Interventions: Drug: Ceftaroline Fosamil; Drug: Ampicillin; Drug: Aminoglycoside

INTERVENTIONS:
Drug: Ceftaroline Fosamil — Ceftaroline fosamil will be given at a dose of 6 mg/kg IV over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour).
  Other Names: Zinforo, Teflaro
Drug: Ampicillin — Ampicillin IV is required for the first 48 hours if the presence of an organism that requires treatment with ampicillin cannot be excluded. Will be given as per local standard of care.
Drug: Aminoglycoside — Optional, will be given as per local standard of care.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ceftaroline for the treatment of Late Onset Sepsis in neonates and young infants aged 7 to <60 days

DETAILED DESCRIPTION:
This is a multicentre, multinational, open-label, single treatment arm study of intravenous (IV) ceftaroline fosamil and ampicillin, plus an optional aminoglycoside of choice, in hospitalized neonates and young infants aged 7 to < 60 days with late-onset sepsis (LOS).

Baseline assessments for study eligibility will occur within 36 hours before administration of the first dose of study therapy. Study Day 1 is defined as the 24-hour period starting at the onset of the first administration of study therapy. Thereafter, subsequent Study Days are to follow the same pattern.

Safety assessments will occur throughout the study. Clinical outcome evaluations will occur at End-of-Therapy (EOT; within 24 hours after completion of last infusion) and Test-of-Cure (TOC; 8 to 15 days after the last dose of study therapy).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent in writing from parent(s) or other legally-acceptable representative(s);
* Male or female, gestational age ≥34 weeks, and chronological age 7 to <60 days at the time of screening;
* Diagnosis of sepsis within 36 hours before enrolment, defined as the presence of at least 2 clinical criteria and at least 1 laboratory criterion in the presence of or as a result of suspected or proven bacterial infection that requires IV antibiotic therapy;
* Patients must meet at least 2 of the following clinical criteria :Hypothermia (<36°C) OR fever (>38.5°C); Bradycardia OR tachycardia OR rhythm instability; Urine output 0.5 to 1 mL/kg/h OR hypotension OR mottled skin OR impaired peripheral perfusion; Petechial rash OR sclerema neonatorum; New onset or worsening of apnoea episodes OR tachypnoea episodes OR increased oxygen requirements OR requirement for ventilation support; Feeding intolerance OR poor sucking OR abdominal distension; Irritability; Lethargy; Hypotonia:
* Patients must meet at least 1 of the following laboratory criteria: White blood cell count ≤4,000 × 109/L OR ≥20,000 × 109/L; Immature to total neutrophil ratio >0.2; Platelet count ≤100,000 × 109/L; C-reactive protein (CRP) >15 mg/L OR procalcitonin ≥2 ng/mL; Hyperglycaemia OR Hypoglycaemia; Metabolic acidosis.

Exclusion Criteria:

* Documented history of any hypersensitivity or allergic reaction to any β-lactam antibiotic or aminoglycoside;
* At study entry, has confirmed infection with a pathogen known to be resistant to the combination of ceftaroline fosamil, ampicillin, and the optional aminoglycoside of choice OR confirmed viral, fungal, or parasitic pathogen as the sole cause of infection;
* Refractory septic shock within 24 hours before enrolment that does not resolve after 60 minutes of vasopressor therapy;
* Moderate or severe renal impairment defined as serum creatinine ≥2 times the upper limit of normal (× ULN) for age OR urine output <0.5 mL/kg/h (measured over at least 8 hours) OR requirement for dialysis;
* Evidence of progressively fatal underlying disease, or life expectancy of ≤60 days;
* Documented history of seizure;
* Requiring or currently taking antiretroviral therapy for human immunodeficiency virus (HIV) or a child from an HIV positive mother;
* Proven or suspected central nervous system (CNS) infection (eg, meningitis, brain abscess, subdural abscess), osteomyelitis, endocarditis, or necrotizing enterocolitis (NEC);
* Any condition (eg, cystic fibrosis, urea cycle disorders), antepartum/peripartum factors, or procedures that would, in the opinion of the investigator, make the patient unsuitable for the study, place a patient at risk, or compromise the quality of data;
* Patient's parent(s) or legally-acceptable representative(s) involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). Concurrent participation in another clinical study with an investigational product (IP), previous enrolment/participation in this study, or participation in another study of ceftaroline fosamil within 14 days before the intended start of the first dose of study therapy.

Ages: 7 Days to 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Rady Children's Hospital San Diego, San Diego, California, United States
- Hungary (3):
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz - Rendelointezet, Gyermekinfektologiai Osztaly, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Gyermek-, Koraszulott es Csecsemoosztaly, Budapest
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Gyermekosztaly, Nyíregyháza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley JS, Stone GG, Chan PLS, Raber SR, Riccobene T, Mas Casullo V, Yan JL, Hendrick VM, Hammond J, Leister-Tebbe HK. Phase 2 Study of the Safety, Pharmacokinetics and Efficacy of Ceftaroline Fosamil in Neonates and Very Young Infants With Late-onset Sepsis. Pediatr Infect Dis J. 2020 May;39(5):411-418. doi: 10.1097/INF.0000000000002607. PMID 32091493
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=D3720C00009&StudyName=Open-label%2C+Multicentre+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+Pharmacokinetics%2C+And+Efficacy+Of+Ceftaroline+In+Neonates+And+Young+Infants+With+Late-onset+Sepsis

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceftaroline Fosamil: Young Infants: Young infants aged greater than (>) 28 days to less than (<) 60 days, received ceftaroline fosamil infusion, intravenously (IV) at a dose of 4 milligrams per kilogram (mg/kg) or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
- Ceftaroline Fosamil: Term Neonates: Term Neonates (defined as gestational age greater than or equal to [>=] 37 weeks) aged 7 to less than equal to (<=28) days received ceftaroline fosamil infusion, IV at a dose of 4 mg/kg or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
- Ceftaroline Fosamil: Preterm Neonates: Preterm neonates (defined as gestational age >=34 weeks to <37 weeks) aged 7 to <=28 days received ceftaroline fosamil infusion, IV at a dose of 4 mg/kg or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
Period: Overall Study
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates
Started | 4 | 5 | 2
Treated | 4 | 5 | 2
Completed | 2 | 3 | 2
Not Completed | 2 | 2 | 0
Not completed — Treatment stopped to be discharged home | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set consisted of all enrolled participants for whom informed consent form was signed.
Groups:
- Ceftaroline Fosamil: Young Infants: Young infants aged >28 days to <60 days, received ceftaroline fosamil infusion, IV at a dose of 4 mg/kg or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
- Ceftaroline Fosamil: Term Neonates: Term Neonates (defined as gestational age >= 37 weeks) aged 7 to <=28 days received ceftaroline fosamil infusion, IV at a dose of 4 mg/kg or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
- Total: Total of all reporting groups
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates | Total
Number analyzed (Participants) | 4 | 5 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: days] | 48.0 (4.69) | 22.0 (3.81) | 15.5 (4.95) | 30.3 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 1 | 4 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 5 | 2 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Discontinuations Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to study follow-up (SFU) visit (28 to 35 days after last dose of study treatment) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to SFU visit (up to a maximum study duration of 49 days)
Population: Safety analysis set consisted of all enrolled participants for whom informed consent form was signed and received any amount of ceftaroline fosamil.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates
Number analyzed (Participants) | 4 | 5 | 2
Participants
  AEs | 1 | 3 | 1
  SAEs | 0 | 0 | 1
  Discontinuations Due to AEs | 0 | 0 | 0

2. Secondary Outcome: Plasma Concentration of Ceftaroline Fosamil
Description: Data was not summarized and provided for individual participants only and reported in this end point for only those participants who had concentrations above limit of quantification (LOQ). LOQ was 50 nanogram per milliliter (ng/mL).
Time Frame: At the end of infusion (EOI)
Population: Pharmacokinetic (PK) analysis set included all participants who received a known amount of ceftaroline fosamil, were randomized to a PK sample collection schedule, and had at least 1 PK sample collected.
Measure: Number; unit: ng/mL
Groups:
- Ceftaroline Fosamil: All Participants: All participants who received ceftaroline fosamil infusion, IV at a dose of 4 mg/kg or 6 mg/kg over 60 minutes every 8 hours in combination with ampicillin IV as per local standard of care, for a minimum of 48 hours and up to a maximum duration of 14 days. Along with this, participants received an aminoglycoside which was optional and could be started and stopped at any time during the study at the discretion of investigator.
Arm/Group | Ceftaroline Fosamil: All Participants
Number analyzed (Participants) | 11
ng/mL
  Participant 1 | 67.7
  Participant 2 | 63.7
  Participant 3 | 74.5

3. Secondary Outcome: Plasma Concentration of Ceftaroline
Description: Ceftaroline fosamil was the prodrug of ceftaroline. Data was not summarized and provided for individual participants only and reported in this end point for only those participants who had concentrations above LOQ at any specific time-point. LOQ was 50 ng/mL
Time Frame: At EOI, 15 minutes to 2 hours, 3 to 4 hours and 5 to 7 hours after EOI
Population: PK analysis set included all participants who received a known amount of ceftaroline fosamil, were randomized to a PK sample collection schedule, and had at least 1 PK sample collected.
Measure: Number; unit: ng/mL
Arm/Group | Ceftaroline Fosamil: All Participants
Number analyzed (Participants) | 11
ng/mL
  Participant 1: 3 to 4 hrs EOI | 3420
  Participant 2: At EOI | 12400
  Participant 2: At 3 to 4 hours after EOI | 4280
  Participant 3: At EOI | 7890
  Participant 3: At 3 to 4 hours after EOI | 1760
  Participant 4: At 15 minutes to 2 hours after EOI | 9440
  Participant 4: At 5 to 7 hours after EOI | 1800
  Participant 5: At EOI | 9410
  Participant 6: 15 minutes to 2 hours after EOI | 4370
  Participant 7: At 15 minutes to 2 hours after EOI | 5550
  Participant 7: At 5 to 7 hours after EOI | 1870
  Participant 8:At 15 minutes to 2 hours after EOI | 2240
  Participant 8: At 5 to 7 hours after EOI | 4770
  Participant 9: At 15 minutes to 2 hours after EOI | 4750
  Participant 9: At 5 to 7 hours after EOI | 1700
  Participant 10: At EOI | 9700
  Participant 10: At 3 to 4 hours after EOI | 3550
  Participant 11: At 15 minutes to 2 hours after EOI | 4760
  Participant 11: At 5 to 7 hours after EOI | 2440

4. Secondary Outcome: Plasma Concentration of Ceftaroline M-1
Description: Ceftaroline M-1 was the inactive metabolite of ceftaroline. Data was not summarized and provided for individual participants only and reported in this end point for only those participants who had concentrations above LOQ at any specific time-point. LOQ was 50 ng/mL
Time Frame: At EOI, 15 minutes to 2 hours, 3 to 4 hours and 5 to 7 hours after EOI
Population: The PK analysis set will include all participants who received a known amount of ceftaroline fosamil, were randomized to a PK sample collection schedule, and had at least 1 PK sample collected.
Measure: Number; unit: ng/mL
Arm/Group | Ceftaroline Fosamil: All Participants
Number analyzed (Participants) | 11
ng/mL
  Participant 1: At 3 to 4 hours after EOI | 729
  Participant 2: At EOI | 678
  Participant 2: At 3 to 4 hours after EOI | 749
  Participant 3: At EOI | 950
  Participant 3: At 3 to 4 hours after EOI | 559
  Participant 4: At 15 minutes to 2 hours after EOI | 970
  Participant 4: At 5 to 7 hours after EOI | 642
  Participant 5: At EOI | 850
  Participant 6: At 15 minutes to 2 hours after EOI | 832
  Participant 7: At 15 minutes to 2 hours after EOI | 728
  Participant 7: At 5 to 7 hours after EOI | 634
  Participant 8: At 15 minutes to 2 hours after EOI | 630
  Participant 8: At 5 to 7 hours after EOI | 785
  Participant 9: At 15 minutes to 2 hours after EOI | 592
  Participant 9: At 5 to 7 hours after EOI | 461
  Participant 10: At EOI | 575
  Participant 10: At 3 to 4 hours after EOI | 648
  Participant 11: At 15 minutes to 2 hours after EOI | 671
  Participant 11: At 5 to 7 hours after EOI | 646

5. Secondary Outcome: Percentage of Participants With Favorable Clinical Response
Description: Clinical response was assessed by the investigator as Cure, Failure or Indeterminate at End of treatment (EOT) and Test of Cure (TOC). Favorable clinical response was defined as clinical response of Cure (defined as resolution of all acute signs and symptoms of Late-onset sepsis [LOS] or improvement to such an extent that no further antibacterial therapy is required). EOT visit occurred within 24 hours after the end of last infusion. TOC visit occurred within 8 to 15 days after the last dose of study therapy.
Time Frame: EOT visit (up to Day 15), TOC visit (up to Day 29)
Population: Modified ITT analysis set: participants who received ceftaroline fosamil and met minimal disease criteria of late-onset sepsis (diagnosis of sepsis within 36 hours before enrolment [defined as presence of >=2 clinical criteria, >=1 laboratory criteria in presence of or as a result of suspected /proven bacterial infection that requires IV therapy]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates
Number analyzed (Participants) | 4 | 3 | 1
percentage of participants
  At EOT visit | 50.0 [12.3 to 87.7] | 33.3 [3.9 to 82.3] | 100 [14.7 to 100]
  At TOC visit | 50.0 [12.3 to 87.7] | 33.3 [3.9 to 82.3] | 100 [14.7 to 100]

6. Secondary Outcome: Percentage of Participants With Favorable Microbiological Response
Description: Microbiological response was determining programmatically and assessed at the participants level at EOT and TOC. Microbiological response was defined as Favorable (Eradication or Presumed Eradication), Unfavorable (Persistence or Presumed Persistence) or Indeterminate (participant's clinical response is Indeterminate and no microbiological culture data is available). Eradication defined as absence of the original baseline pathogen from the source specimen; presumed eradication was defined when source specimen was not available to culture and the participant was assessed as a clinical cure (resolution of all acute signs and symptoms of LOS or improvement to such an extent that no further antibacterial therapy was required). EOT visit occurred within 24 hours after the end of last infusion. TOC visit occurred within 8 to 15 days after last dose of study drug.
Time Frame: EOT visit (up to Day 15), TOC visit (up to Day 29)
Population: Modified ITT analysis set: participants who received ceftaroline fosamil and met minimal disease criteria of late-onset sepsis (diagnosis of sepsis within 36 hours before enrolment [defined as presence of >=2 clinical criteria, >=1 laboratory criteria in presence of or as a result of suspected /proven bacterial infection that requires IV therapy).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates
Number analyzed (Participants) | 4 | 3 | 1
percentage of participants
  At EOT visit | 50.0 [12.3 to 87.7] | 66.7 [17.7 to 96.1] | 100 [14.7 to 100]
  At TOC visit | 25.0 [2.8 to 71.6] | 33.3 [3.9 to 82.3] | 100 [14.7 to 100]

ADVERSE EVENTS:
Time Frame: Baseline up to SFU visit (up to a maximum study duration of 49 days)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Ceftaroline Fosamil: Young Infants | Ceftaroline Fosamil: Term Neonates | Ceftaroline Fosamil: Preterm Neonates
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 1/2
Other Adverse Events (participants affected / at risk) | 1/4 | 3/5 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftaroline Fosamil: Young Infants (N=4) | Ceftaroline Fosamil: Term Neonates (N=5) | Ceftaroline Fosamil: Preterm Neonates (N=2)
Salmonellosis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftaroline Fosamil: Young Infants (N=4) | Ceftaroline Fosamil: Term Neonates (N=5) | Ceftaroline Fosamil: Preterm Neonates (N=2)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0
Rhinitis (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT02424734/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02424734/SAP_001.pdf